CLINICAL TRIAL: NCT01303107
Title: A Non-Inferiority Phase 3 Comparative Study Between a Heavy Levobupivacaine in 50% Enantiomeric Excess (Bupivacaine S75:R25) and Heavy Racemic Bupivacaine for Cesarean Operation
Brief Title: Comparative Mixture of Non-racemic and Racemic Enantiomers of Bupivacaine in Cesarean
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor has no interest in continuing the study.
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Irmandade da Santa Casa da Misericórdia de Santos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CRIST019
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2011-01

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine S50:R50 (Active Comparator): 3 ml subarachnoid block
  Interventions: Drug: Bupivacaine
- bupivacaine S75:R25 (Experimental): 3 ml for subarachnoid block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — single dose of 15 mg by a slow injection rate of 1 mL/s
  Other Names: Marcaine

SUMMARY:
The purpose of this study is to determine if the mixture of enantiomers of bupivacaine (bupivacaine S75:R25) dos not represent inferiority efficacy and safety compare to the racemic mixture of enantiomers of bupivacaine (bupivacaine S50:R50).

DETAILED DESCRIPTION:
The enantiomeric mixture of bupivacaine S75:R25 (75% levobupivacaine and 25% bupivacaine) was develop to be a safety regional anesthetic in substitution to racemic bupivacaine (S50:R50).

ELIGIBILITY:
Inclusion Criteria:

* parturients at term
* ASA (American Society of Anesthesiologists) I or ASA II
* elective cesarean section with low risk labor
* pre-natal follow-up
* patient consent

Exclusion Criteria:

* relative or absolute contraindications for spinal anesthesia
* history of hypersensitivity to the local anesthetics
* use of opioids during labor
* labor lasting more than 12 hours or less than 1 hour
* complications of pregnancy such as placenta previa, pre-eclampsia or eclampsia; maternal-fetal malnutrition;important accidents during pregnancy.
* spinal lesions, peripheral neuropathies or any other neurologic disorders that lead to changes of sensitivity and/or motricity
* decompensated diabetes or hypertension
* history of alcohol and/or drug abuse
* cardiopathies, especially myocardiopathies and valvulopathies; important cognitive changes
* changes in safety exams
* twin pregnancy;
* signs of intrauterine distress, and abnormalities of fetal vitality, prematurity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
latency of sensitive block at T6 | loss of pain in T6
  The anesthesiologist will evaluate the loss of pain to pin-prick in T10.

SECONDARY OUTCOMES:
duration of the anesthesia | recovery of the sensibility
  Time to recover the sensibility due to the anesthetic
Degree of motor block | End of motor block
  Evaluated by the Bromage scale after the injection of the anesthetic solution
maximal level of the sensitive blockade | last level of sensitive blockade
  Evaluation by pin-prick every 2 minutes after the injection of the anesthetic solution.
Maternal cardiocirculatory and respiratory parameters | During the study
  systolic and diastolic blood pressure (SBP and DBP), heart rate (HR), and oxygen saturation (SpO2) are evaluate during the study
Parturients ambulation | regression of the motor blockade
  Will be measured the time that the parturients ambulate, due to de regression of the motor blockade
Visceral pain | suture of the peritoneum
  Visceral pain will be assessed at the time of suture of the peritoneum.
Neonatal repercussions | birth of the neonatal
  Evaluation of the Apgar index in the first and fifth minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Liga Mathias, PhD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (2):
- Brazil (2):
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos, São Paulo
  - Irmandade da Santa Casa de Misericóridia de São Paulo, São Paulo, São Paulo